CLINICAL TRIAL: NCT07159360
Title: Safety, Usability, and Effectiveness of a Gait Exoskeleton for Children and Adolescents With Neurodevelopmental Disorders.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); APAC, I.A.P. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXC
Record Dates: First submitted 2025-05-23; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Neuromuscular Disorders; Neurodevelopmental Disorders
Keywords: Neurodevelopmental disorders; Neuromuscular disorders; cerebral palsy; acquired brain injury; spinal muscular atrophy; robotics; gait; spinal cord injury
MeSH Terms: conditions — Neuromuscular Diseases; Neurodevelopmental Disorders; Cerebral Palsy; Brain Injuries; Muscular Atrophy, Spinal; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLINICAL EXPLORER (Experimental): An initial assessment (screening visit), 8 intervention sessions (2 per week) in the rehabilitation center, and a final assessment.
  Interventions: Device: CLINICAL EXPLORER

INTERVENTIONS:
Device: CLINICAL EXPLORER — 8 sessions of use of the device in the rehabilitation center

SUMMARY:
Neurodevelopmental disorders often result in abnormal development of the Central Nervous System (CNS), frequently causing motor dysfunctions such as the inability to stand and walk. CLINICAL EXPLORER is a clinical-use robotic device for gait training, representing the evolution of the ATLAS 2030 exoskeleton and the EXPLORER device for home use. The aim of this study is to evaluate the safety and usability of CLINICAL EXPLORER .

DETAILED DESCRIPTION:
Neuromuscular and neurological disorders in children cause muscle weakness and spasticity, leading to severe motor dysfunctions such as the inability to maintain posture or walk. Manually assisted gait training can be physically demanding for therapists, which is why robotic devices have been developed to reduce their workload, provide objective assessments through integrated sensors, and improve rehabilitation quality. Beyond mobilizing muscles and joints, these devices enhance brain neuroplasticity and the child's connectivity with their environment, positively impacting self-esteem and social interaction. A clinical-use robotic device for gait training has been developed, representing the evolution of the ATLAS 2030 exoskeleton and the EXPLORER device for home use.

ELIGIBILITY:
Inclusion Criteria for Phase 0

* Age between 2 and 17 years.
* Consent from the participant or legal guardian to participate in the study.
* No diagnosis of neurodevelopmental disorders such as CP, NMD, LM, or MS. Inclusion Criteria for Phase 1
* Age between 2 and 17 years.
* Consent from the participant or legal guardian to participate in the study.
* Diagnosis of neurodevelopmental disorders such as CP, NMD, LM, or MS. Inclusion Criteria Related to the EXPLORER CLINICAL Device Characteristics
* Medical authorization to stand upright and perform weight-bearing gait training.
* Weight less than or equal to 60 kg.
* Hip width less than or equal to 40 cm.
* Distance from the hip joint center to the knee joint center: 21 cm - 36 cm.
* Distance from the knee joint center to the ankle joint center: 20 - 35 cm.
* EU shoe size less than or equal to 40.

Exclusion Criteria:

* Any medical contraindication for standing or walking.
* Presence of non-reducible contractures or heterotopic ossification above the degrees allowed by the device and/or outside the trajectory imposed by the device.
* Spasticity (MAS) = 4 in lower limbs at the time of device use.
* Structured hip and/or knee contracture greater than 20 degrees.
* Inability to stand or walk with more than 5 degrees of hip abduction.
* Inability to achieve 5 degrees of dorsal ankle flexion from the neutral position with or without orthosis.
* Tibial leg length discrepancy that cannot be mitigated with the use of a foot wedge.
* Skin alterations in areas of contact with the device.
* History of fracture without trauma.
* Presence of other conditions that cause exercise intolerance (such as uncontrolled hypertension, coronary artery diseases, arrhythmia, congestive heart failure, severe pulmonary disease).
* Behavioral disorders that interfere with proper use of the device, such as impulsivity.
* Allergy to any of the materials of the EXPLORER CLÍNICO: cotton, nylon, polyester, PPS, PEEK, or ABS. The materials used in EXPLORER CLÍNICO that were not previously used in ATLAS 2030, a medical device certified by the AEMPS, are PPS, PEEK, and ABS.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | through study completion, along 8 weeks
  occurrence of any serious adverse event to the participant or the caregiver
Falls prevalence | through study completion, along 8 weeks
  Number of falling events occurred from the participant or caregiver
Skin integrity | through study completion, along 8 weeks
  Occurrence of any injury of the skin in the areas of contact and produced by the use of the device
Pain (Visual Analogic Scale) | through study completion, along 8 weeks
  pain measured by the Visual Analogic Scale (VAS) by the participant and the caregiver, scored from 0 to 10, being 0 "no pain" and 10 "unbearable pain"
Heart rate | through study completion, along 8 weeks
  measurement of heart rate with a smart band
Oxygen saturation | through study completion, along 8 weeks
  measurement of Oxygen saturation with a smart band
Blood pressure | through study completion, along 8 weeks
  measurement of blood pressure with a smart band
Donning and doffing time | through study completion, along 8 weeks
  Time to don and doff the device to each participant
QUEST | at the end of the intervention at 8 weeks
  Using the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) questionnaire administered to the participants' caregivers at the end of the intervention. The QUEST 2.0 scale has 12 items. Each item is rated on a 5-point Likert scale

SECONDARY OUTCOMES:
Gait analysis | Day 1 and at the end of the intervention at 8 weeks
  Spatiotemporal parameters will be done through photogrammetry.
Range of motion | Day 1 and at the end of the intervention at 8 weeks
  Passive Degree to which a joint can move (hip, knee, and ankle joints in both legs). From 0º to 180º.
Quality of life (EQ-5D) | Day 1 and at the end of the intervention at 8 weeks
  The EQ-5D is a standardized instrument used to measure and evaluate the quality of life. It assesses five key dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 3-level or 5-level scale, reflecting the severity of the condition (e.g., no problems, some problems, or extreme problems). The EQ-5D also includes a visual analogue scale (VAS) where individuals rate their overall health on a scale from 0 to 100. The tool is widely used in clinical trials, health surveys, and economic evaluations to assess health-related quality of life and make comparisons across different patient populations or interventions.
Level of fatigue | through study completion, along 8 weeks
  Fatigue of both the participant and the therapist, Measured with the Borg scale
Level of Spasticity | Day 1 and through study completion, along 8 weeks
  Evaluation of spasticity with Modified Ahsworth Scale
Muscular activity (EMG) | through study completion, along 8 weeks
  EMG (Electromyography) is a technique that measures the electrical activity of muscles to assess their function. It helps detect neuromuscular disorders and evaluate muscle activation patterns, using either surface electrodes or needle inserts to record muscle activity. Measured with the system FREEEMG/BTS®.
Cerebral activity (EEG) | through study completion, along 8 weeks
  EEG (Electroencephalography) is a method used to record electrical activity in the brain. It involves placing electrodes on the scalp to measure brain wave patterns, helping to diagnose conditions like epilepsy, sleep disorders, and brain injuries. Measured with Enobio® EEG systems.
Acceptability | at the end of the intervention, 8th week
  Analysis of the drop-out rate during the study period
Accessibility of the participant | through study completion, along 8 weeks
  Rate of the participants suitable to use the device

CONTACTS AND LOCATIONS:
Locations (2):
- Asociación Pro Personas con Paralisis Cerebral (APAC-IAP), Mexico City, Mexico City, Mexico
- Hospital Infantil Universitario Niño Jesús-Servicio de Neuro Ortopedia, Madrid, Madrid, Spain